CLINICAL TRIAL: NCT03403270
Title: Testing the Efficacy of the ENCOURAGE App in Decreasing Sedentary Behaviour: A Time Series Quasi-Experimental Study
Brief Title: A Mobile Health App to Reduce Sedentary Time in Inactive Employees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Boniface Hospital (Other)
Collaborators: Heart and Stroke Foundation Manitoba (Unknown); Tactica Interactive Winnipeg (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H2016:228
Record Dates: First submitted 2017-10-12; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Physical Activity; Sedentary Lifestyle
Keywords: Mobile App; Sedentary Behaviour; Workplace Wellness; Sitting Time
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Time Series Quasi-Experiment
Masking Description: Outcome Assessors will not be aware of previous research data collected. As this is a single group study, all participants will receive the intervention as described.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ENCOURAGE App Intervention (Experimental): Users will download the ENCOURAGE mobile app. The App uses a time management technique (i.e. Pomodoro technique) as a strategy to provide prompts for users to engage in an activity. The App can be customized by the users to set prompts at intervals that fit into their schedule. For example, these activities can range from a stretching activity (e.g., a neck stretch), a standing activity (e.g., stand and read), or a physical activity (e.g., fill up the printer with paper, do a squat). Additionally, the App will use Behaviour Change Techniques as a strategy to support participants as they reduce their sedentary behaviour and improve their physical activity levels. The App uses a series of Behavior Change Techniques shown to be effective in promoting a more active lifestyle.
  Interventions: Other: ENCOURAGE App

INTERVENTIONS:
Other: ENCOURAGE App — Users will have an opportunity to engage with the app as described for the duration of the study period.

SUMMARY:
The ENCOURAGE App will use mobile health technology to support employees to reduce their sedentary time and become more physically active. The mobile app has been developed using time management techniques (i.e. Pomodoro technique) as a strategy to provide prompts to encourage users to engage in an activity and break up bouts of prolonged sitting.

DETAILED DESCRIPTION:
Sixty percent of Canadian adults are accessible through the workplace. Thus, workplace wellness programs that include physical activity components provide a viable option to encourage employees to reduce sedentary time. Moving forward with the ENCOURAGE health promotion model, we will use mobile health technology to support employees to reduce sitting and become more physically active, while offering employers a solution that can be easily implemented in a variety of contexts.

The public release of the ENCOURAGE App will involve two phases:

1. The recruitment of up to 300 individuals through the App. Any user will be able to download the ENCOURAGE App through the iTunes Store or Google Play. Note that when participants download the App, they are not automatically enrolled in the study. Participants will be prompted, after downloading the App, with a brief description of the study, as well as a pre-screening tool that will be used to determine eligibility. Users will be asked via a pop-up to determine if they wish to participate in a research project. Users will be asked to participate in a time series quasi-experimental study to determine if the ENCOURAGE App can support participants to increase the number of breaks in sedentary time taken throughout the day, over a 6-month time period. The App can be customized by the users to set prompts at intervals that fit into their schedule. For example, these activities can range from a stretching activity (e.g., a neck stretch), a standing activity (e.g., stand and read), or a physical activity (e.g., fill up the printer with paper, do a squat). Additionally, the App will use Behaviour Change Techniques as a strategy to support participants as they reduce their sedentary behaviour and increase their physical activity levels.
2. The recruitment of a sub-sample of 60 participants who live in Winnipeg, MB which will be drawn from the larger sample. In addition to completing all the components of the larger research study, the sub-sample will be also asked to wear a physical activity monitor, called an accelerometer.

The objectives of this study are to determine if the final product ENCOURAGE App:

1. Reduces the number of breaks from sitting;
2. Reduces total sedentary time;
3. Increases physical activity levels; and,
4. Improves self-efficacy for reducing sedentary behaviour.

ELIGIBILITY:
Inclusion Criteria:

-Specific to sub-sample of 60 participants; live in Winnipeg, MB

Exclusion Criteria:

* Individuals who do not own a personal mobile phone
* Any physical limitations that would not allow individual to engage in physical activity
* Any cognitive limitations that would not allow individual to consent for study
* Specific to sub-sample of 60 participants; live outside Winnipeg, MB

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-01-31 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of breaks from sitting | Change from baseline number of breaks from sitting at 1-month
  This outcome will be assessed by self-report using the Workplace Sitting Breaks Questionnaire.

SECONDARY OUTCOMES:
Number of breaks from sitting | Change from baseline number of breaks from sitting at 1-week, 2-months, 3-months, 4-months, 5-months, and 6-months
  This outcome will be assessed by self-report using the Workplace Sitting Breaks Questionnaire in a typical work day
Duration of breaks from sitting | Change from baseline duration of breaks from sitting at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  This outcome will be assessed by self-report using the Workplace Sitting Breaks in a typical work day.
Percent time spent sitting at work | Change from baseline percent time spent sitting at work at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  This outcome will be assessed by the Occupational Sitting and Physical Activity Questionnaire over the last 7 days
Percent time spent standing at work | Change from baseline percent time spent standing at work at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  This outcome will be assessed by the Occupational Sitting and Physical Activity Questionnaire over the last 7 days
Percent time spent walking at work | Change from baseline percent time spent walking at work at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  This outcome will be assessed by the Occupational Sitting and Physical Activity Questionnaire over the last 7 days
Percent time spent participating in heavy labour at work | Change from baseline percent time spent participating in heavy labour at work at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  This outcome will be assessed by the Occupational Sitting and Physical Activity over the last 7 days
Mild physical activity | Change from baseline minutes per week in mild physical activity at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  This outcome will be assessed by the Godin Leisure-Time Exercise Questionnaire in minutes per week
Moderate physical activity | Change from baseline minutes per week in moderate physical activity at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  This outcome will be assessed by the Godin Leisure-Time Exercise Questionnaire in minutes per week
Strenuous physical activity | Change from baseline minutes per week in strenuous physical activity at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  This outcome will be assessed by the Godin Leisure-Time Exercise Questionnaire in minutes per week
Degree of confidence to break up sitting time | Change from baseline degree of confidence to break up sitting time at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  This outcome will be assessed by the Task Self-Efficacy for Sedentary Behaviour Questionnaire using a scale from 0 (i.e. not at all confident) to 10 (i.e. completely confident)
Degree of confidence for engaging in self-regulatory actions that would help them reduce their sedentary time | Change from baseline degree of confidence for engaging in self-regulatory actions that would help them reduce their sedentary time at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  This outcome will be assessed by the Self-Regulatory Efficacy for Sedentary Behaviour Questionnaire using a scale from 0 (i.e. not at all confident) to 10 (i.e. completely confident)
Degree of confidence for reducing their sedentary behaviours even when faced with feeling tired at work | Change from baseline for reducing their sedentary behaviours even when faced with feeling tired at work at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  This outcome will be assessed by the Self-Regulatory Efficacy for Managing Barriers Questionnaire using a scale from 10 (i.e. not at all confident) to 100 (i.e. completely confident)
Degree of confidence for reducing their sedentary behaviours even when faced with feeling comfortable in their seated position at work | Change from baseline for reducing their sedentary behaviours even when faced with feeling comfortable in their seated position at work at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  This outcome will be assessed by the Self-Regulatory Efficacy for Managing Barriers Questionnaire using a scale from 10 (i.e. not at all confident) to 100 (i.e. completely confident)
Degree of confidence for reducing their sedentary behaviours even when having important tasks to do while seated at work | Change from baseline for reducing their sedentary behaviours even when having important tasks to do while seated at work at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  This outcome will be assessed by the Self-Regulatory Efficacy for Managing Barriers Questionnaire using a scale from 10 (i.e. not at all confident) to 100 (i.e. completely confident)
Degree of confidence for reducing their sedentary behaviours even when feeling as if they deserve to sit at work | Change from baseline for reducing their sedentary behaviours even when feeling as if they deserve to sit at work at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  This outcome will be assessed by the Self-Regulatory Efficacy for Managing Barriers Questionnaire using a scale from 10 (i.e. not at all confident) to 100 (i.e. completely confident)
Degree of confidence for reducing their sedentary behaviours even when feeling stressed at work | Change from baseline for reducing their sedentary behaviours even when feeling stressed at work at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  This outcome will be assessed by the Self-Regulatory Efficacy for Managing Barriers Questionnaire using a scale from 10 (i.e. not at all confident) to 100 (i.e. completely confident)
Degree of confidence for reducing their sedentary behaviours even when feeling down or depressed at work | Change from baseline for reducing their sedentary behaviours even when feeling down or depressed at work at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  This outcome will be assessed by the Self-Regulatory Efficacy for Managing Barriers Questionnaire using a scale from 10 (i.e. not at all confident) to 100 (i.e. completely confident)
Total sedentary time | Change from baseline total sedentary time at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  Sub-sample of 60 individuals will wear an accelerometer to measure their total sedentary time (hours per day)
Prolonged bouts of sedentary time lasting at least 30 minutes | Change from baseline prolonged bouts of sedentary time lasting at least 30 minutes at 1-week, 1-month, 2-month, 3-month, 4-month, 5-month, 6-month
  Sub-sample of 60 individuals will wear an accelerometer to measure their prolonged bouts of sedentary time lasting at least 30 minutes (number per day)

CONTACTS AND LOCATIONS:
Locations (1):
- St-Boniface Hospital Albrechtsen Research Center, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
We do not intend to share individual participant data with researchers outside of the principal and co-investigators.

REFERENCES:
- [Background] Stamatakis E, Hamer M, Dunstan DW. Screen-based entertainment time, all-cause mortality, and cardiovascular events: population-based study with ongoing mortality and hospital events follow-up. J Am Coll Cardiol. 2011 Jan 18;57(3):292-9. doi: 10.1016/j.jacc.2010.05.065. PMID 21232666
- [Background] Dunstan DW, Barr EL, Healy GN, Salmon J, Shaw JE, Balkau B, Magliano DJ, Cameron AJ, Zimmet PZ, Owen N. Television viewing time and mortality: the Australian Diabetes, Obesity and Lifestyle Study (AusDiab). Circulation. 2010 Jan 26;121(3):384-91. doi: 10.1161/CIRCULATIONAHA.109.894824. Epub 2010 Jan 11. PMID 20065160
- [Background] Wilmot EG, Edwardson CL, Achana FA, Davies MJ, Gorely T, Gray LJ, Khunti K, Yates T, Biddle SJ. Sedentary time in adults and the association with diabetes, cardiovascular disease and death: systematic review and meta-analysis. Diabetologia. 2012 Nov;55(11):2895-905. doi: 10.1007/s00125-012-2677-z. Epub 2012 Aug 14. PMID 22890825
- [Background] Thorp AA, Owen N, Neuhaus M, Dunstan DW. Sedentary behaviors and subsequent health outcomes in adults a systematic review of longitudinal studies, 1996-2011. Am J Prev Med. 2011 Aug;41(2):207-15. doi: 10.1016/j.amepre.2011.05.004. PMID 21767729
- [Background] Proper KI, Singh AS, van Mechelen W, Chinapaw MJ. Sedentary behaviors and health outcomes among adults: a systematic review of prospective studies. Am J Prev Med. 2011 Feb;40(2):174-82. doi: 10.1016/j.amepre.2010.10.015. PMID 21238866
- [Background] van Uffelen JG, Wong J, Chau JY, van der Ploeg HP, Riphagen I, Gilson ND, Burton NW, Healy GN, Thorp AA, Clark BK, Gardiner PA, Dunstan DW, Bauman A, Owen N, Brown WJ. Occupational sitting and health risks: a systematic review. Am J Prev Med. 2010 Oct;39(4):379-88. doi: 10.1016/j.amepre.2010.05.024. PMID 20837291
- [Background] Colley RC, Garriguet D, Janssen I, Craig CL, Clarke J, Tremblay MS. Physical activity of Canadian adults: accelerometer results from the 2007 to 2009 Canadian Health Measures Survey. Health Rep. 2011 Mar;22(1):7-14. PMID 21510585
- [Background] Thorp AA, Healy GN, Winkler E, Clark BK, Gardiner PA, Owen N, Dunstan DW. Prolonged sedentary time and physical activity in workplace and non-work contexts: a cross-sectional study of office, customer service and call centre employees. Int J Behav Nutr Phys Act. 2012 Oct 26;9:128. doi: 10.1186/1479-5868-9-128. PMID 23101767
- [Background] Tew GA, Posso MC, Arundel CE, McDaid CM. Systematic review: height-adjustable workstations to reduce sedentary behaviour in office-based workers. Occup Med (Lond). 2015 Jul;65(5):357-66. doi: 10.1093/occmed/kqv044. Epub 2015 May 1. PMID 25934982
- [Background] Neuhaus M, Healy GN, Dunstan DW, Owen N, Eakin EG. Workplace sitting and height-adjustable workstations: a randomized controlled trial. Am J Prev Med. 2014 Jan;46(1):30-40. doi: 10.1016/j.amepre.2013.09.009. PMID 24355669
- [Background] Evans RE, Fawole HO, Sheriff SA, Dall PM, Grant PM, Ryan CG. Point-of-choice prompts to reduce sitting time at work: a randomized trial. Am J Prev Med. 2012 Sep;43(3):293-7. doi: 10.1016/j.amepre.2012.05.010. PMID 22898122
- [Background] Shrestha N, Kukkonen-Harjula KT, Verbeek JH, Ijaz S, Hermans V, Bhaumik S. Workplace interventions for reducing sitting at work. Cochrane Database Syst Rev. 2016 Mar 17;3(3):CD010912. doi: 10.1002/14651858.CD010912.pub3. PMID 26984326
- [Background] Verweij LM, Proper KI, Weel AN, Hulshof CT, van Mechelen W. The application of an occupational health guideline reduces sedentary behaviour and increases fruit intake at work: results from an RCT. Occup Environ Med. 2012 Jul;69(7):500-7. doi: 10.1136/oemed-2011-100377. Epub 2012 Mar 1. PMID 22383591
- [Background] Allen JC, Lewis JB, Tagliaferro AR. Cost-effectiveness of health risk reduction after lifestyle education in the small workplace. Prev Chronic Dis. 2012;9:E96. doi: 10.5888/pcd9.110169. Epub 2012 May 10. PMID 22575081
- [Background] Free C, Phillips G, Galli L, Watson L, Felix L, Edwards P, Patel V, Haines A. The effectiveness of mobile-health technology-based health behaviour change or disease management interventions for health care consumers: a systematic review. PLoS Med. 2013;10(1):e1001362. doi: 10.1371/journal.pmed.1001362. Epub 2013 Jan 15. PMID 23349621
- [Background] Hurling R, Catt M, Boni MD, Fairley BW, Hurst T, Murray P, Richardson A, Sodhi JS. Using internet and mobile phone technology to deliver an automated physical activity program: randomized controlled trial. J Med Internet Res. 2007 Apr 27;9(2):e7. doi: 10.2196/jmir.9.2.e7. PMID 17478409
- [Background] Stephens J, Allen J. Mobile phone interventions to increase physical activity and reduce weight: a systematic review. J Cardiovasc Nurs. 2013 Jul-Aug;28(4):320-9. doi: 10.1097/JCN.0b013e318250a3e7. PMID 22635061
- [Background] Fanning J, Mullen SP, McAuley E. Increasing physical activity with mobile devices: a meta-analysis. J Med Internet Res. 2012 Nov 21;14(6):e161. doi: 10.2196/jmir.2171. PMID 23171838
- [Background] Abraham C, Michie S. A taxonomy of behavior change techniques used in interventions. Health Psychol. 2008 May;27(3):379-87. doi: 10.1037/0278-6133.27.3.379. PMID 18624603
- [Background] Michie S, Richardson M, Johnston M, Abraham C, Francis J, Hardeman W, Eccles MP, Cane J, Wood CE. The behavior change technique taxonomy (v1) of 93 hierarchically clustered techniques: building an international consensus for the reporting of behavior change interventions. Ann Behav Med. 2013 Aug;46(1):81-95. doi: 10.1007/s12160-013-9486-6. PMID 23512568
- [Background] Mohr DC, Cheung K, Schueller SM, Hendricks Brown C, Duan N. Continuous evaluation of evolving behavioral intervention technologies. Am J Prev Med. 2013 Oct;45(4):517-23. doi: 10.1016/j.amepre.2013.06.006. PMID 24050429
- [Background] Collins LM, Murphy SA, Strecher V. The multiphase optimization strategy (MOST) and the sequential multiple assignment randomized trial (SMART): new methods for more potent eHealth interventions. Am J Prev Med. 2007 May;32(5 Suppl):S112-8. doi: 10.1016/j.amepre.2007.01.022. PMID 17466815
- [Background] Kumar S, Nilsen WJ, Abernethy A, Atienza A, Patrick K, Pavel M, Riley WT, Shar A, Spring B, Spruijt-Metz D, Hedeker D, Honavar V, Kravitz R, Lefebvre RC, Mohr DC, Murphy SA, Quinn C, Shusterman V, Swendeman D. Mobile health technology evaluation: the mHealth evidence workshop. Am J Prev Med. 2013 Aug;45(2):228-36. doi: 10.1016/j.amepre.2013.03.017. PMID 23867031
- [Background] Williams SL, French DP. What are the most effective intervention techniques for changing physical activity self-efficacy and physical activity behaviour--and are they the same? Health Educ Res. 2011 Apr;26(2):308-22. doi: 10.1093/her/cyr005. Epub 2011 Feb 14. PMID 21321008
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Eysenbach G; CONSORT-EHEALTH Group. CONSORT-EHEALTH: improving and standardizing evaluation reports of Web-based and mobile health interventions. J Med Internet Res. 2011 Dec 31;13(4):e126. doi: 10.2196/jmir.1923. PMID 22209829
- [Background] Prochaska JO, DiClemente CC. Stages and processes of self-change of smoking: toward an integrative model of change. J Consult Clin Psychol. 1983 Jun;51(3):390-5. doi: 10.1037//0022-006x.51.3.390. No abstract available. PMID 6863699
- [Background] Michie S, Ashford S, Sniehotta FF, Dombrowski SU, Bishop A, French DP. A refined taxonomy of behaviour change techniques to help people change their physical activity and healthy eating behaviours: the CALO-RE taxonomy. Psychol Health. 2011 Nov;26(11):1479-98. doi: 10.1080/08870446.2010.540664. Epub 2011 Jun 28. PMID 21678185
- [Background] Pedisic Z, Bennie JA, Timperio AF, Crawford DA, Dunstan DW, Bauman AE, Salmon J. Workplace Sitting Breaks Questionnaire (SITBRQ): an assessment of concurrent validity and test-retest reliability. BMC Public Health. 2014 Dec 5;14:1249. doi: 10.1186/1471-2458-14-1249. PMID 25476788
- [Background] Maclagan LC, Park J, Sanmartin C, Mathur KR, Roth D, Manuel DG, Gershon A, Booth GL, Bhatia S, Atzema CL, Tu JV. The CANHEART health index: a tool for monitoring the cardiovascular health of the Canadian population. CMAJ. 2014 Feb 18;186(3):180-7. doi: 10.1503/cmaj.131358. Epub 2013 Dec 23. PMID 24366893
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Blumenthal JA. Depression and coronary heart disease: association and implications for treatment. Cleve Clin J Med. 2008 Mar;75 Suppl 2:S48-53. doi: 10.3949/ccjm.75.suppl_2.s48. PMID 18540147
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Chau JY, Van Der Ploeg HP, Dunn S, Kurko J, Bauman AE. Validity of the occupational sitting and physical activity questionnaire. Med Sci Sports Exerc. 2012 Jan;44(1):118-25. doi: 10.1249/MSS.0b013e3182251060. PMID 21659903
- [Background] Rothney MP, Schaefer EV, Neumann MM, Choi L, Chen KY. Validity of physical activity intensity predictions by ActiGraph, Actical, and RT3 accelerometers. Obesity (Silver Spring). 2008 Aug;16(8):1946-52. doi: 10.1038/oby.2008.279. Epub 2008 May 29. PMID 18535553
- [Background] Colley RC, Tremblay MS. Moderate and vigorous physical activity intensity cut-points for the Actical accelerometer. J Sports Sci. 2011 May;29(8):783-9. doi: 10.1080/02640414.2011.557744. PMID 21424979
- [Background] Welk GJ, Schaben JA, Morrow JR Jr. Reliability of accelerometry-based activity monitors: a generalizability study. Med Sci Sports Exerc. 2004 Sep;36(9):1637-45. PMID 15354049
- [Background] Holmen H, Torbjornsen A, Wahl AK, Jenum AK, Smastuen MC, Arsand E, Ribu L. A Mobile Health Intervention for Self-Management and Lifestyle Change for Persons With Type 2 Diabetes, Part 2: One-Year Results From the Norwegian Randomized Controlled Trial RENEWING HEALTH. JMIR Mhealth Uhealth. 2014 Dec 11;2(4):e57. doi: 10.2196/mhealth.3882. PMID 25499872
- [Background] Kannisto KA, Korhonen J, Adams CE, Koivunen MH, Vahlberg T, Valimaki MA. Factors Associated With Dropout During Recruitment and Follow-Up Periods of a mHealth-Based Randomized Controlled Trial for Mobile.Net to Encourage Treatment Adherence for People With Serious Mental Health Problems. J Med Internet Res. 2017 Feb 21;19(2):e46. doi: 10.2196/jmir.6417. PMID 28223262
- [Background] Fukuoka Y, Gay C, Haskell W, Arai S, Vittinghoff E. Identifying Factors Associated With Dropout During Prerandomization Run-in Period From an mHealth Physical Activity Education Study: The mPED Trial. JMIR Mhealth Uhealth. 2015 Apr 13;3(2):e34. doi: 10.2196/mhealth.3928. PMID 25872754

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT03403270/SAP_000.pdf
  • Study Protocol (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT03403270/Prot_001.pdf